CLINICAL TRIAL: NCT03142087
Title: The Effect of Virtual Reality Exercises on Balance in Children With Brain Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Müberra TANRIVERDİ, lecturer, PT, MSc, PhD (c), Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mtanriverdi88
Record Dates: First submitted 2017-03-31; First posted 2017-05-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Postural Balance
Keywords: balance; brain tumor; virtual reality
MeSH Terms: conditions — Brain Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality exercises (Active Comparator): Nintendo Wii Fit Plus Game Console is used in these group. The one session included:warm-up exercises in 5-10 minutes, games (soccer heading, ski jump, ski slalom, etc.) in 30-40 minutes, and cooling exercises in 5 minutes.
  Interventions: Other: exercises
- conventional exercises (Active Comparator): Physiotherapy and rehabilitation session included: warm-up exercises in 5-10 minutes, balance exercises (balance board, balance ball, two and one leg stand exercises, weight bearing exercises, balance in different type of surfaces, etc.) in 30-40 minutes, and cooling exercises in 5 minutes.
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — exercise

SUMMARY:
30 patients with brain tumor will be included in the study between the ages of 6 and 18 who have undergone surgery. Patients included in the study will be randomly assigned to two groups. The study group will be included in the Nintendo Wii Fit Plus Balance Game exercise program under the supervision of a physiotherapist for 2 days per week for 8 weeks. The control group will be taken to the conventional exercise program under the supervision of a physiotherapist for 2 days a week, 1 hour a day. The assessments will be made before the exercise program begins and at the end of the 8th week. Patients' physical measurements were assessed by anthropometric evaluations, muscle strength measurement, pain Visual Analogue Scale, walking Observational Walking Analysis, Balanced Pediatric Functional Range Test, Timed Up and Go (TUG) and one foot standing test and Nintendo Wii Fit Plus Balance Assessment, Functional capacity 2 min. With Walking Test, fatigue with PedsQL Multidimensional Fatigue Scale, daily life activities will be evaluated with WeeFIM.

DETAILED DESCRIPTION:
In our pediatric rehabilitation policlinic we have seen that these children has problems in balance and coordination from cause muscle weakness and cerebral-sensory-proprioceptive problems. We have evaluated with all parameters belong the physiotherapy and rehabilitation measurements and then planning this study with study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 years of children
* brain tumor

Exclusion Criteria:

* have any conditions with exercises
* neurological and musculoskeletal disorders

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
the effects of virtual reality exercises evaluating with Nintendo Wii Fit Plus on balance | change from baseline balance at 8 weeks
  Nintendo Wii Fit Plus Game Console evaluation parameters which are percentage of weight bearing and central of gravity

CONTACTS AND LOCATIONS:
Overall Officials: Müberra Tanrıverdi, PT, MSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided